CLINICAL TRIAL: NCT02761265
Title: The Effect of Thoracolumbar Spinal Deformity and Its Surgical Correction on Gait and Balance in Adults
Brief Title: Gait and Balance in Thoracolumbar Spinal Deformity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Back Institute (Other)
Collaborators: Alphatec Spine, Inc. (Industry)
Responsible Party: Principal Investigator, Ram Haddas, Director of Research, Texas Back Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TBIRF-SBL-003
Record Dates: First submitted 2016-04-19; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Spinal Curvatures
Keywords: Degenerative Adult Scoliosis; Gait Analysis; Balance Analysis; Biomechanics; Neuromuscular Control; Thoracolumbar Deformity
MeSH Terms: conditions — Spinal Curvatures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical Group (Experimental): Gait and balance testing as well as self-reported outcome assessments to be administered before and after surgery
  Interventions: Procedure: Surgical intervention
- Control Group (Other): Gait and balance testing to be administered once in healthy subjects
  Interventions: Other: None (Asymptomatic group)

INTERVENTIONS:
Procedure: Surgical intervention — Surgery to correct spinal deformity
  Arms: Surgical Group
Other: None (Asymptomatic group) — Gait and balance testing performed, no treatment in this asymptomatic group
  Arms: Control Group

SUMMARY:
Surgical intervention may provide pain relief and improvement in function but one area of significant clinical interest is the restoration/improvement in gait and functional balance. Based on the investigators knowledge, there is limited literature on biomechanics and neuromuscular control of the lower extremities and spine as assessed by objective gait analysis and balance strategies in adult degenerative scoliosis patients, pre and post surgical intervention. The purpose of this study is to determine the impact of spinal deformity on the biomechanics and neuromuscular control of the lower and upper extremities, and also investigate the impact of surgery on these functions as evaluated by gait and balance analyses using dynamic EMG, video motion capture and force plate analysis and also to compare these patients with healthy controls to better evaluate the extent of limitations before and after surgery.

DETAILED DESCRIPTION:
Degenerative adult scoliosis results from age related changes leading to segmental instability, deformity and stenosis. Although the etiology is unclear, degenerative adult scoliosis is associated with progressive and asymmetric degeneration of the disc and facet joints, which typically lead to stenosis. By virtue of the narrowed spinal canal associated with the degeneration these patients frequently develop back pain, as well as leg pain, weakness, and numbness. With an aging population in the USA and an increased attention to quality of life versus cost issues in the current healthcare environment, degenerative adult scoliosis has become a considerable healthcare concern.

Patients with scoliosis demonstrate an altered gait pattern. Such differences include decreased step length and reduced range of motion in the upper and lower extremities, asymmetry of trunk rotation and ground reaction force in three-dimensions. Mahaudens et al. found a decrease in the muscular mechanical work associated with an increase of energy cost and a decrease in the muscular efficiency in a scoliosis population compared to healthy controls. Furthermore, scoliosis patients exert 30% more physical effort than healthy subjects to ensure habitual locomotion, and this additional effort requires a reciprocal increase of oxygen consumption. This altered gait pattern demonstrated by subjects with scoliosis may be due to changes in global postural control strategies caused by spinal deformity.

Previous research showed that scoliosis patients do not have impaired postural balance when compared to healthy controls, while several others did find an effect of scoliosis on postural balance. This discrepancy in findings may be due to differences in curve characteristics included and their effects on postural balance, curve types (single or double), number of different curve types, location of curves (thoracic and lumbar), and/or Cobb angles. Furthermore, Schimmel et al. found that postural balance one year after surgery did not improve as a result of the better spinal alignment, neither did the reduced range of trunk motion inherent to fusion negatively affect postural balance.

While medicinal interventions may assist with some of the associated co-morbid conditions, surgical interventions may be indicated for those patients with intractable and debilitating low back and leg pain. These surgeries have proven to be extremely successful in a majority of patients. The surgeries may involve decompression and instrumentation to stabilize the spine to achieve arthrodesis.

Surgical intervention may provide pain relief and improvement in function but one area of significant clinical interest is the restoration/improvement in gait and functional balance. Based on the investigators knowledge, there is limited literature on biomechanics and neuromuscular control of the lower extremities and spine as assessed by objective gait analysis and balance strategies in adult degenerative scoliosis patients, pre and post surgical intervention. The purpose of this study is to determine the impact of spinal deformity on the biomechanics and neuromuscular control of the lower and upper extremities, and also investigate the impact of surgery on these functions as evaluated by gait and balance analyses using dynamic Electromyograph (EMG), video motion capture and force plate analysis and also to compare these patients with healthy controls to better evaluate the extent of limitations before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 years and older
2. Clinically diagnosed thoracolumbar and/or lumbo-sacro-pelvic deformity as defined by the SRS/Schwab classification systems as Cobb angle of 25° or greater
3. Instrumentation to be used at 4 or more levels
4. Able to ambulate without assistance and stand without assistance with participant eyes open for a minimum of 10 seconds
5. Able and willing to attend and perform the activities described in the informed consent within the boundaries of the timelines set forth for pre-, and post-operative follow-up

Exclusion Criteria:

1. History of prior attempt at fusion (successful or not) at the indicated levels, (history of one level fusion is not an exclusion)
2. Major lower extremity surgery or previous injury that may affect gait (a successful total joint replacement is not an exclusion)
3. BMI higher than 35
4. Neurological disorder, diabetic neuropathy or other disease that impairs the patient's ability to ambulate or stand without assistance
5. Usage of blood thinners
6. Major trauma to the pelvis
7. Pregnant or wishing to become pregnant during the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Kinematic Variables Change assessed with human motion capture system | Prior to surgery; 3 and 12 months after surgery
  3-Dimensional Range of Motion (ROM) during the stance and swing phase.
Kinetic Variables Change assessed with human motion capture system | Prior to surgery; 3 and 12 months after surgery
  Vertical Ground Reaction Forces (GRF)
Electromyography Variables Change assessed with an Electromyograph | Prior to surgery; 3 and 12 months after surgery
  Bilateral peak magnitude during the stance phase
Spatio-Temporal Variables Change assessed with human motion capture system | Prior to surgery; 3 and 12 months after surgery
  Walking Speed

SECONDARY OUTCOMES:
Patient Self-Reported Outcome Assessments Change | Prior to surgery; 3 and 12 months after surgery
  Visual Analog Scale (VAS)
Patient Self-Reported Outcome Assessments Change | Prior to surgery; 3 and 12 months after surgery
  Scoliosis Research Society (SRS) -22
Patient Self-Reported Outcome Assessments Change | Prior to surgery; 3 and 12 months after surgery
  Neck Disability Index (NDI)
Patient Self-Reported Outcome Assessments Change | Prior to surgery; 3 and 12 months after surgery
  Oswestry Disability Index (ODI)

CONTACTS AND LOCATIONS:
Overall Officials: Ram Haddas, PhD, Principal Investigator — Texas Back Institute
Locations (1):
- Texas Back Institute, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotwal S, Pumberger M, Hughes A, Girardi F. Degenerative scoliosis: a review. HSS J. 2011 Oct;7(3):257-64. doi: 10.1007/s11420-011-9204-5. Epub 2011 Jun 11. PMID 23024623
- [Background] Kotwicki T, Chowanska J, Kinel E, Czaprowski D, Tomaszewski M, Janusz P. Optimal management of idiopathic scoliosis in adolescence. Adolesc Health Med Ther. 2013 Jul 23;4:59-73. doi: 10.2147/AHMT.S32088. eCollection 2013. PMID 24600296
- [Background] Ploumis A, Transfledt EE, Denis F. Degenerative lumbar scoliosis associated with spinal stenosis. Spine J. 2007 Jul-Aug;7(4):428-36. doi: 10.1016/j.spinee.2006.07.015. Epub 2007 Feb 28. PMID 17630141
- [Background] Engsberg JR, Bridwell KH, Reitenbach AK, Uhrich ML, Baldus C, Blanke K, Lenke LG. Preoperative gait comparisons between adults undergoing long spinal deformity fusion surgery (thoracic to L4, L5, or sacrum) and controls. Spine (Phila Pa 1976). 2001 Sep 15;26(18):2020-8. doi: 10.1097/00007632-200109150-00016. PMID 11547203
- [Background] Yang JH, Suh SW, Sung PS, Park WH. Asymmetrical gait in adolescents with idiopathic scoliosis. Eur Spine J. 2013 Nov;22(11):2407-13. doi: 10.1007/s00586-013-2845-y. Epub 2013 Jun 4. PMID 23732766
- [Background] Mahaudens P, Banse X, Mousny M, Detrembleur C. Gait in adolescent idiopathic scoliosis: kinematics and electromyographic analysis. Eur Spine J. 2009 Apr;18(4):512-21. doi: 10.1007/s00586-009-0899-7. Epub 2009 Feb 18. PMID 19224255
- [Background] Arima H, Yamato Y, Hasegawa T, et al. Gait analysis after corrective surgery for adult spinal deformity - good sagittal balance with improved lumber lordosis is important. Scoliosis. 2015;10(Suppl 1):O76.
- [Background] Kramers-de Quervain IA, Muller R, Stacoff A, Grob D, Stussi E. Gait analysis in patients with idiopathic scoliosis. Eur Spine J. 2004 Aug;13(5):449-56. doi: 10.1007/s00586-003-0588-x. Epub 2004 Apr 3. PMID 15064994
- [Background] Schizas CG, Kramers-de Quervain IA, Stussi E, Grob D. Gait asymmetries in patients with idiopathic scoliosis using vertical forces measurement only. Eur Spine J. 1998;7(2):95-8. doi: 10.1007/s005860050037. PMID 9629931
- [Background] Chockalingam N, Dangerfield PH, Rahmatalla A, Ahmed el-N, Cochrane T. Assessment of ground reaction force during scoliotic gait. Eur Spine J. 2004 Dec;13(8):750-4. doi: 10.1007/s00586-004-0762-9. Epub 2004 Jun 22. PMID 15221574
- [Background] Giakas G, Baltzopoulos V, Dangerfield PH, Dorgan JC, Dalmira S. Comparison of gait patterns between healthy and scoliotic patients using time and frequency domain analysis of ground reaction forces. Spine (Phila Pa 1976). 1996 Oct 1;21(19):2235-42. doi: 10.1097/00007632-199610010-00011. PMID 8902968
- [Background] Mahaudens P, Detrembleur C, Mousny M, Banse X. Gait in adolescent idiopathic scoliosis: energy cost analysis. Eur Spine J. 2009 Aug;18(8):1160-8. doi: 10.1007/s00586-009-1002-0. Epub 2009 Apr 24. PMID 19390877
- [Background] O'Beirne J, Goldberg C, Dowling FE, Fogarty EE. Equilibrial dysfunction in scoliosis--cause or effect? J Spinal Disord. 1989 Sep;2(3):184-9. PMID 2520074
- [Background] Kuo FC, Wang NH, Hong CZ. Impact of visual and somatosensory deprivation on dynamic balance in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2010 Nov 1;35(23):2084-90. doi: 10.1097/BRS.0b013e3181cc8108. PMID 20975488
- [Background] Karimi MT, Kavyani M, Kamali M. Balance and gait performance of scoliotic subjects: A review of the literature. J Back Musculoskelet Rehabil. 2016 Aug 10;29(3):403-15. doi: 10.3233/BMR-150641. PMID 26519115
- [Background] Beaulieu M, Toulotte C, Gatto L, Rivard CH, Teasdale N, Simoneau M, Allard P. Postural imbalance in non-treated adolescent idiopathic scoliosis at different periods of progression. Eur Spine J. 2009 Jan;18(1):38-44. doi: 10.1007/s00586-008-0831-6. Epub 2008 Dec 6. PMID 19066989
- [Background] Schimmel JJ, Groen BE, Weerdesteyn V, de Kleuver M. Adolescent idiopathic scoliosis and spinal fusion do not substantially impact on postural balance. Scoliosis. 2015 Jun 9;10:18. doi: 10.1186/s13013-015-0042-y. eCollection 2015. PMID 26056528
- [Background] Guo X, Chau WW, Hui-Chan CW, Cheung CS, Tsang WW, Cheng JC. Balance control in adolescents with idiopathic scoliosis and disturbed somatosensory function. Spine (Phila Pa 1976). 2006 Jun 15;31(14):E437-40. doi: 10.1097/01.brs.0000222048.47010.bf. PMID 16778672
- [Background] Simoneau M, Mercier P, Blouin J, Allard P, Teasdale N. Altered sensory-weighting mechanisms is observed in adolescents with idiopathic scoliosis. BMC Neurosci. 2006 Oct 19;7:68. doi: 10.1186/1471-2202-7-68. PMID 17052338
- [Background] Sachs D, Capobianco R, Cher D, Holt T, Gundanna M, Graven T, Shamie AN, Cummings J Jr. One-year outcomes after minimally invasive sacroiliac joint fusion with a series of triangular implants: a multicenter, patient-level analysis. Med Devices (Auckl). 2014 Aug 28;7:299-304. doi: 10.2147/MDER.S56491. eCollection 2014. PMID 25210479
- [Background] Toosizadeh N, Yen TC, Howe C, Dohm M, Mohler J, Najafi B. Gait behaviors as an objective surgical outcome in low back disorders: A systematic review. Clin Biomech (Bristol). 2015 Jul;30(6):528-36. doi: 10.1016/j.clinbiomech.2015.04.005. Epub 2015 Apr 17. PMID 25921552
- [Background] Portney LG, Watkins MP. Foundation of clinical research: applications to practice. 3rd ed. Upper Saddle River, New Jersy: Julie Levin Alexander; 2009.
- [Background] Schwab F, Ungar B, Blondel B, Buchowski J, Coe J, Deinlein D, DeWald C, Mehdian H, Shaffrey C, Tribus C, Lafage V. Scoliosis Research Society-Schwab adult spinal deformity classification: a validation study. Spine (Phila Pa 1976). 2012 May 20;37(12):1077-82. doi: 10.1097/BRS.0b013e31823e15e2. PMID 22045006
- [Background] El Fegoun AB, Schwab F, Gamez L, Champain N, Skalli W, Farcy JP. Center of gravity and radiographic posture analysis: a preliminary review of adult volunteers and adult patients affected by scoliosis. Spine (Phila Pa 1976). 2005 Jul 1;30(13):1535-40. doi: 10.1097/01.brs.0000167534.49069.e9. PMID 15990669
- [Background] Vaughan CL, Davis BL, O'Conner JC. Dynamics of Human Gait. 2nd ed. Cape Town, South Africa: Kiboho Publishers; 1999.
- [Background] Arumugam A, Milosavljevic S, Woodley S, Sole G. Effects of external pelvic compression on form closure, force closure, and neuromotor control of the lumbopelvic spine--a systematic review. Man Ther. 2012 Aug;17(4):275-84. doi: 10.1016/j.math.2012.01.010. Epub 2012 Mar 2. PMID 22386280